CLINICAL TRIAL: NCT00152373
Title: A Double-blind, Placebo-controlled, Randomized Study: 16-week Evaluation of the Efficacy and Safety of Levetiracetam (LEV) as add-on Therapy in Adults and Adolescents Older Than 16 Years Suffering From Partial Seizures.
Brief Title: Double-blind, Placebo-controlled Study of Levetiracetam in Adults With POS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: N01102
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy, Partial Onset Seizures; Keppra; Levetiracetam
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
clinical efficacy and safety of Levetiracetam as add-on therapy in adult Chinese subjects with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

1. subject suffering from partial onset seizures, whether or not secondarily generalized,
2. presence of the following during the eight weeks of the historical baseline period: at least eight partial seizures (type IA, IB or IC) with or without secondary generalization.
3. subject on a stable dose of at least one and no more than two other concomitant antiepileptic drugs (AEDs).
4. subject who has been exposed to at least one classical AEDs,
5. CT scan or MRI performed within the last 2 years and free of neoplasia, progressive cerebral disease or any other progressively neurodegenerative disease.

Exclusion Criteria:

1. history of status epilepticus within three months prior to the Selection visit,
2. subjects whose seizures cannot reliably be counted on a regular basis due to their fast and repetitive occurrence (clusters or flurries),
3. use of any medication (other than the concomitant AED) that influences the central nervous system (CNS) unless on a stable regimen for at least 1 month prior to the Selection visit. Antidepressants (except amitriptyline, mianserin and fluoxetine), anxiolytics and hypnotics are allowed. Intermittent benzodiazepines are allowed as long as the frequency is not greater than one single administration per week for at least 3 months prior to the Selection visit. Neuroleptics and Traditional Chinese AEDs are not allowed.,
4. history or presence of pseudoseizures,

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 192
Dates: Start 2004-07; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The partial onset (type I) seizure frequency reduction per week over the 16-week treatment period (titration and maintenance)

SECONDARY OUTCOMES:
Seizure freedom ;
The partial onset (type I) seizure reduction response rate ;
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma